CLINICAL TRIAL: NCT00214591
Title: A 52-wk Randomised, Double-Blind, Parallel-Group, Multi-Centre, Active-Controlled (Metformin) Study to Evaluate the Efficacy, Safety & Tolerability of Tesaglitazar Therapy When Administered to Patients With Type 2 Diabetes
Brief Title: GALLANT 5 Tesaglitazar Versus Metformin
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The development program has been terminated
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D6160C00029
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — tesaglitazar

INTERVENTIONS:
Drug: GALIDA

SUMMARY:
This is a 52-week randomized, double-blind, parallel-group, multi-center, active-controlled (metformin) study of tesaglitazar in patients with type 2 diabetes, not adequately controlled on diet and lifestyle advice alone during the run-in period. The study comprises a 6 week placebo single blind run in period followed by a 52-week a double blind treatment period and a 3-week follow-up period. Tesaglitazar and metformin will be titrated to optimal effect or highest tolerable dose during the first 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Provision of a written informed consent
* Men or women who are ³18 years of age
* Female patients: postmenopausal, hysterectomized, or if of childbearing potential, using a reliable method of birth control
* Diagnosed with type 2 diabetes
* Treated with diet alone or treatment with a single oral antidiabetic agent or low doses of two oral antidiabetic agents

Exclusion Criteria:

* Type 1 diabetes
* New York Heart Association heart failure Class III or IV
* Treatment with chronic insulin
* History of hypersensitivity or intolerance to any peroxisome proliferator-activated receptor agonist (like Actos or Avandia), fenofibrate, metformin or 3-hydroxy-3-methylglutaryl coenzyme A reductase inhibitor (statin)
* History of drug-induced myopathy or drug-induced creatine kinase elevation, liver enzyme elevations, neutropenia (low white blood cells)
* Creatinine levels above twice the normal range
* Creatine kinase above 3 times the upper limit of normal
* Received any investigational product in other clinical studies within 12 weeks
* Any clinically significant abnormality identified on physical examination, laboratory tests or electrocardiogram, which in the judgment of the investigator would compromise the patient's safety or successful participation in the clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580
Dates: Start 2004-08; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Absolute change from baseline to end of randomized treatment period in glycosylated hemoglobin A1c (HbA1c)

SECONDARY OUTCOMES:
The change in fasting plasma glucose (FPG), insulin, proinsulin and C-peptide
Insulin sensitivity by assessment of change in the calculated variable homeostasis assessment model
Lipid parameters (triglyceride [TG], total cholesterol, high-density lipoprotein cholesterol [HDL C], non-HDL C, low-density lipoprotein cholesterol [LDL C], apolipoproteins [Apo] A-I, Apo B, Apo CIII, free fatty acids, lipoprotein particle size and co
C-reactive protein, LDL C/HDL C ratio and Apo B/Apo A-I ratio
FPG, homeostasis assessment model, insulin, proinsulin, C-peptide
Tumor necrosis factor-alpha, intracellular adhesion molecule-1
Fibrinogen
Urinary albumin excretion
Waist/hip ratio
Responder analyses for HbA1c, FPG, TG, HDL C, total cholesterol, non HDL C and LDL C according to pre-specified values
Proportion of patients reaching pre-specified target levels for HbA1c, FPG, TG, HDL C, non-HDL C and LDL C
Pharmacokinetics of tesaglitazar
Safety and tolerability of tesaglitazar by assessment of adverse events, laboratory values, electrocardiogram, pulse, blood pressure, hypoglycemic events, body weight, cardiac evaluation, and physical examination

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Galida Medical Science Director, MD, Study Director — AstraZeneca
Locations (130):
- United States (64):
  - Research Site, Birmingham, Alabama
  - Research Site, Columbiana, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Carlisle, Arizona
  - Research Center, Sherwood, Arizona
  - Research Site, Chula Vista, California
  - Research Site, Escondido, California
  - Research Site, Huntington Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Mission Viejo, California
  - Research Site, Orange, California
  - Research Site, Pasadena, California
  - Research Site, Pomona, California
  - Research Site, Redondo Beach, California
  - Research Site, Sacramento, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Wheat Ridge, Colorado
  - Research Site, Clearwater, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Brunswick, Georgia
  - Research Site, Carollton, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Boise, Idaho
  - Research Site, Evansville, Indiana
  - Research Site, Kansas City, Kansas
  - Research Site, Overland Park, Kansas
  - Research Site, Witchita, Kansas
  - Research Site, Bossier City, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Kalamazoo, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Hamilton, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Albany, New York
  - Research Site, New York, New York
  - Research Site, Pahrump, New York
  - Research Site, Rochester, New York
  - Research Site, The Bronx, New York
  - Research Site, White Plains, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Kettering, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Simpsonville, South Carolina
  - Research Site, Morristown, Tennessee
  - Research Site, Corpus Christi, Texas
  - Research Site, Dallas, Texas
  - Research Site, Lubbock, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Burke, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Tacoma, Washington
  - Research Site, Menomonee Falls, Wisconsin
  - Research Site, Milwaukee, Wisconsin
- Finland (10):
  - Research Site, Hämeenlinna
  - Research Site, Helsinki
  - Research Site, Joensuu
  - Research Site, Kouvola
  - Research Site, Kuopio
  - Research Site, Mikkeli
  - Research Site, Oulu
  - Research Site, Salo
  - Research Site, Tampere
  - Research Site, Vantaa
- Germany (18):
  - Research Site, Aschaffenburg
  - Research Site, Bad Segeberg
  - Research Site, Beckum
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Ehrenberg
  - Research Site, Essen
  - Research Site, Feldafing
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Hermaringen
  - Research Site, Künzing
  - Research Site, Langen
  - Research Site, Mannheim
  - Research Site, Marl
  - Research Site, Nuremberg
  - Research Site, Pirna
  - Research Site, Rotenburg/Fulda
- Israel (7):
  - Research Site, Ashkelon
  - Research Site, Haifa
  - Research Site, Holon
  - Research Site, Jerusalem
  - Research Site, Rishon LeZiyyon
  - Research Site, Safed
  - Research Site, Tel Aviv
- Netherlands (10):
  - Research Site, Beek en Donk
  - Research Site, Bennebroe
  - Research Site, Deurne
  - Research Site, Huizen
  - Research Site, Losser
  - Research Site, Nijverdal
  - Research Site, Rijswijk
  - Research Site, Roelofarendsveen
  - Research Site, Rotterdam
  - Research Site, The Hague
- Norway (3):
  - Research Site, Bergen
  - Research Site, Oslo
  - Research Site, Østerås
- Spain (7):
  - Research Site, San Vicente de Raspeig, Alicante
  - Research Site, Villar del Arzobispo, Valencia
  - Research Site, Alzira (Valencia)
  - Research Site, Barcelona
  - Research Site, Begonte (Lugo)
  - Research Site, Madrid
  - Research Site, Seville
- United Kingdom (11):
  - Research Site, Aberdeen
  - Research Site, Ayr
  - Research Site, Bath
  - Research Site, Berks
  - Research Site, Bucks
  - Research Site, Coventry
  - Research Site, Dundee
  - Research Site, Glasgow
  - Research Site, Manchester
  - Research Sites, Northampton
  - Research Site, Wiltshire